CLINICAL TRIAL: NCT03271333
Title: Description of the Functional Evolution of Diffuse Infiltrating Pneumonia Associated With Systemic Scleroderma and Analysis of Associated Factors.
Brief Title: Description of the Functional Evolution of Diffuse Infiltrating Pneumonia Associated With Systemic Scleroderma.
Acronym: SCLERO-PID
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2015_49; 2016-A00722-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with systemic sclerosis
  Interventions: Other: lung function tests

INTERVENTIONS:
Other: lung function tests — Patients hospitalized realise a Resting pulmonary function tests (PFT) which include the assessment of ventilatory capacity: spirometry (forced expiratory flows and mobilisable volumes)

SUMMARY:
Diffuse infiltrating pneumonia (DIP) is a severe complication of systemic sclerosis and one of the leading cause of death in this condition. The main objective of this study is to prospectively describe the evolution of DIP overtime and to find prognosis factors.

ELIGIBILITY:
Inclusion Criteria:

* systemic sclerosis
* Diffuse Infiltrating Pneumonia

Exclusion Criteria:

* infection
* other lung diseases
* non French native

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic sclerosis and Diffuse Infiltrating Pneumonia
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
composite criteria: forced vital capacity and CO diffusing capacity | At 24 months
  Degradation of forced vital capacity (FVC) ≥10% and / or DLCO ≥15% of initial values at prospective follow-up at 24 months.

SECONDARY OUTCOMES:
composite criteria: forced vital capacity and CO diffusing capacity | At 12 months
  Degradation of forced vital capacity (FVC) ≥10% and / or DLCO ≥15% of initial values at prospective follow-up at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: David Launay, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Hôpital Claude Huriez, CHU, Lille
  - AH-HP, Hôpital Saint Antoine, Paris

IPD SHARING:
Plan to Share IPD: No